CLINICAL TRIAL: NCT06727448
Title: Translation and Validation of the French Version of the Sleep Regularity Questionnaire: a New Tool to Address the the Challenge of Sleep Health
Acronym: PRIMO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/13
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Chronic Insomnia Disorder; Circadian Rhythm Disorders
Keywords: circadian rhythm disorder; Sleep Regularity Questionnaire; SRQ; chronic insomnia disorder
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: French patients indicated for 14-day actimetry for chronic insomnia or circadian rhythm disorders
  Interventions: Other: SRQ questionnaire

INTERVENTIONS:
Other: SRQ questionnaire — SRQ questionnaire administered at inclusion visit and 14 days after inclusion

SUMMARY:
Sleep is an essential function for physical and mental health. The mismatch between biological rhythms and the social rhythms of individuals is increasingly common in modern societies. This sleep irregularity can have numerous consequences on mental health, cardiometabolic health, the immune system, functioning, and quality of life. To address the public health issue of sleep irregularity, it is important to be able to obtain a valid and reliable measure. The Sleep Regularity Questionnaire (SRQ) by Dzierzewski et al. addresses this issue, but has never been translated into French. The aim of the study is to translate and validate the French version of the Sleep Regularity Questionnaire.

DETAILED DESCRIPTION:
Sleep is an essential function for physical and mental health. It involves an interaction between homeostatic regulation (need for sleep in the event of deprivation) and circadian regulation (need for sleep according to day-night alternation). Democratized at the end of the 19th century, electric lighting made nocturnal activities possible, and hence the mismatch between individuals' biological and social rhythms (mismatch of rhythms, sleep irregularity, also known as social jetlag). This sleep irregularity is all the more alarming as it is growing epidemically in our societies, and can have numerous consequences on mental health (anxiety, depression), cardiometabolic health (insulin resistance), the immune system (repeated infections), functioning (driving, cognitive performance), and quality of life. To address the public health issue of sleep irregularity, it is important to be able to obtain a valid and reliable measure. The Sleep Regularity Questionnaire (SRQ) by Dzierzewski et al. addresses this health issue, but has never been translated into French.

The investigators make the following assumptions:

* Cronbach's alpha = 0.87 as in the English version.
* a two-dimensional structure with a circadian regularity factor and a sleep continuity regularity factor will be confirmed by confirmatory factor analyses.
* Convergent validity between SRQ results and actimetric measures of sleep regularity (Sleep Regularity Index, intra-individual variability).

The main objective of this study was to translate and validate the French version of the Sleep Regularity Questionnaire (SRQ).

The secondary objectives are to analyze the external validity (convergent and divergent) of the SRQ by calculating :

* associations with sleep complaints (insomnia, somnolence),
* mental health complaints (depression, anxiety),
* sleep behaviors and electroencephalographic parameters (sleep architecture, fragmentation).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Patient with indication for 14-day actimetry for chronic insomnia or circadian rhythm disorder
* Patients with an indication for 14-day actimetry to assess sleep-wake rhythms, for example prior to a 36-hour polysomnographic recording to diagnose central hypersomnia (narcolepsy or idiopathic hypersomnia).
* Patient affiliated to or benefiting from a social security scheme
* Patient with French as mother tongue, able to read and write French.
* Patient able to understand and complete questionnaires independently
* Patient informed and not opposed to participating in the study

Exclusion Criteria:

* Current psychiatric disorder (mood disorders, anxiety, psychosis, sleep-interfering use disorder) assessed during interview with investigator
* Current neurological disorder affecting sleep (neurodegenerative disease, stroke, epilepsy) assessed during interview with investigator
* Unstable cardiovascular or respiratory diseases
* Pregnant or breast-feeding women
* Adults under guardianship or curatorship
* Opposition to participation expressed by healthy patient/volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French patients indicated for 14-day actimetry for chronic insomnia or circadian rhythm disorders
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Internal validity | At day 14 after inclusion
  consistency measured by Cronbach's alpha and exploratory and confirmatory factor analysis

SECONDARY OUTCOMES:
Insomnia | at inclusion (day 0)
  measured by the Insomnia Severity Index
Sleepiness | at inclusion (day 0)
  measured by the Epworth Sleepiness Scale
Depression and anxiety | at inclusion (day 0)
  measured by the Patient Health Questionnaire-4
Chronotype | at inclusion (day 0)
  measured by the Morningness-Eveningness Scale Short Version
Sleep duration | at inclusion (day 0) and 14 days after inclusion
  measured by actimetry : this examination is used to determine the presence or absence of circadian rhythm disorders and to assess sleep duration s It is the reference examination
Total sleep time | at inclusion (day 0)
  measured by polysomnography

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France